CLINICAL TRIAL: NCT00041990
Title: A Phase II, Multicenter Study of Decitabine (5-Aza-2'Deoxycytidine) in Chronic Myelogenous Leukemia Accelerated Phase Refractory to Imatinib Mesylate (STI 571)
Brief Title: Phase II Trial of Decitabine in Patients With Chronic Myelogenous Leukemia Accelerated Phase Who Are Refractory to Imatinib Mesylate (Gleevec)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Collaborators: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAC-013; DACO-013
Record Dates: First submitted 2002-07-19; First posted 2002-07-23 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic myelogenous leukemia; CML; CML-AP; Accelerated phase; Decitabine; 5-aza-2'deoxycytidine; Methylation; STI 571; Imatinib mesylate; Gleevec; BCR/ABL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine (5-aza-2'deoxycytidine)

SUMMARY:
To determine the safety and efficacy of decitabine in patients with Philadelphia chromosome-positive chronic myelogenous leukemia accelerated phase that were previously treated with imatinib mesylate (STI 571) and became resistant/refractory or were found to be intolerant to the drug.

ELIGIBILITY:
Inclusion:

* Histologically confirmed diagnosis of CML accelerated phase
* Ph chromosome-positive
* Previous treatment with imatinib mesylate resulting in:

  i) Hematologic Resistance / Hematologic Refractory: Based on a physician's (documented) decision to discontinue imatinib mesylate treatment due to failure of continued benefit or no benefit to the patient, ii) Imatinib Mesylate Intolerance: any toxicity resulting in a physician's (documented) decision to discontinue imatinib mesylate treatment.
* Patients must have recovered from the side effects of previous CML therapy for accelerated phase with the exception of hydroxyurea
* Age >/= 2 years
* Bilirubin </= 3 x the upper limit of normal (ULN), SGOT and SGPT </= 3 x ULN, except </= 5 x ULN in leukemic involvement of the liver, serum creatinine </= 2 x ULN
* WHO performance status 0-3
* A negative serum hCG pregnancy test in patients of childbearing potential
* Able to give signed informed consent directly or through a parent or guardian for minors

Exclusion:

* Leukemic involvement of the central nervous system
* Active malignancy other than CML or non-melanoma cancer of the skin
* Previous treatment for CML with another investigational agent within 28 days of study entry
* At study entry, patients who were treated with: imatinib mesylate within the past 48 hours; interferon-alpha within the past 48 hours; homoharringtonine within the past 14 days; low-dose cytosine arabinoside within 7 days, moderate dose within 14 days, or high dose within 28 days; etoposide, anthracyclines, or mitoxantrone within 21 days; busulfan within the past six weeks
* Patients who had received hematopoietic stem cell transplantation within 6 weeks of Day 1 decitabine therapy
* Patients with Grade 3/4 cardiac disease or any other serious concurrent medical condition.
* Patients who are pregnant or nursing. All patients of childbearing potential must practice effective methods of contraception while on study.
* Patients with mental illness or other condition precluding their ability to give informed consent or to comply with study requirements
* Patients with systemic, uncontrolled infections

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - City of Hope Medical Center, Duarte, California
  - Scripps Clinic, Escondido, California
  - USC/Norris Cancer Center, Los Angeles, California
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - New York Medical College, Valhalla, New York
  - Liberty Hematology/Oncology, Columbia, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada